CLINICAL TRIAL: NCT02759952
Title: Clinical Characterization on PDE6A-related Retinitis Pigmentosa in Preparation to a Gene Therapy Trial: An Observational Study
Brief Title: Clinical Characterization on PDE6A-related Retinitis Pigmentosa in Preparation to a Gene Therapy Trial
Status: Completed | Type: Observational
Sponsor: STZ eyetrial (Other)
Responsible Party: Sponsor
Other Study IDs: RDC-PDE6A-00
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; PDE6A; gene therapy trial
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (DNA) for genetic validation of genotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mutations in the PDE6A gene - encoding the -subunit of the rod cGMP-phosphodiesterase - account for 1% of autosomal recessive retinitis pigmentosa (arRP) through impaired regulation of cGMP levels in the rod outer segment. This study aims for a detailed clinical characterization of patients with PDE6A mutations in preparation of a clinical gene replacement study (phase I/II safety trial).

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a clinically and genetically heterogenous group of hereditary retinal disorders, being one of the most common types of retinal degenerations with a prevalence of 1:4000. More than 45 genes have been associated with RP so far, whose defects cause a progressive loss of rod photoreceptor function, followed by cone photoreceptor dysfunction often leading to complete blindness. Mutations in the PDE6A gene - encoding the -subunit of the rod cGMP-phosphodiesterase - account for 1% of autosomal recessive retinitis pigmentosa (arRP) through impaired regulation of cGMP levels in the rod outer segment.

With the help of improved genetic and functional diagnostic tools an early recognition and differentiation has become possible. Still, up to date no established therapy is available, therefore, social and professional consequences are essential tasks to deal with. The modern ophthalmological functional diagnostic tools enable a precise characterisation and early recognition of such retinal diseases. The detailed results and information can help to extend the understanding of the pathological mechanisms involved in these diseases.

In this study the investigators intend to investigate patients with a genetically confirmed diagnosis of Retinitis pigmentosa due to PDE6A mutations hereby assessing the function and structure of the retina with an extensive battery of tests.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis pigmentosa patients with genetically confirmed mutations in the PDE6A-gene
* written informed consent

Exclusion Criteria:

* severe general disease, that would make longer examinations not possible
* patients who cannot give written informed consent independently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinitis pigmentosa patients with genetically confirmed mutations in the PDE6A-gene
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2025-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity in both eyes | 3 years
kinetic visual field in both eyes | 3 years
central retinal thickness in both eyes | 3 years

SECONDARY OUTCOMES:
multifocal ERG responses in both eyes | 3 years
colour vision in both eyes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ditta Zobor, MD, PhD, Principal Investigator — Institute for Ophthalmic Research, University Tübingen, Germany; Susanne Kohl, PhD, Principal Investigator — Institute for Ophthalmic Research, University Tübingen, Germany
Locations (1):
- Institute for Ophthalmic Research, University Tübingen, Germany, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No